CLINICAL TRIAL: NCT05553535
Title: Diagnostic of Rotator Cuff Calcific Tendinosis Using MRI With ZTE Sequence
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, GILLET Romain, MD, Central Hospital, Nancy, France
Other Study IDs: N°1-RCB/EUDRACT
Record Dates: First submitted 2022-09-19; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Cuff Rotator Tendinitis
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: cases of rotator cuff calcific tendinosis on imaging studies
  Interventions: Diagnostic Test: MRI
- witnesses: differential diagnosis or normal cases
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — retrospective review of shoulder MRI

SUMMARY:
Conventional radiographs are still considered the reference for identifying rotator cuff calcific tendinosis.

MRI is widely performed for rotator cuff disorders evaluation but has a moderate accuracy in rotator cuff calcific tendinosis diagnosis and calcific deposits identification (sensitivity and specificity around 60%), even though it helps in determining acuity of the finding by adjacent soft tissue edema depiction and differential diagnosis identification (i.e. adhesive capsulitis, sub-acromial bursitis…).

Zero echo time (ZTE) MRI provides enhanced bone contrast by enabling the acquisition of signals from tissues exhibiting the shortest T2 values on a single sequence with a spatial resolution of 0.8-1.2 mm isotropic and can therefore provide images similar to those obtained with radiographs.

We hypothesize that ZTE images could also depict rotator cuff calcific tendinosis, but to our knowledge, no study compared this technique to radiographs and/or standard MRI.

ELIGIBILITY:
Inclusion Criteria:

* patient referred to the imaging department for a MRI scan in case of suspicion of rotator cuff tendinosis

Exclusion Criteria:

* incomplete data sets

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients over 18 years old referred to our department for a suspicion of rotator cuff tendinosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
calcific deposits presence | Retrospective review of all MRI scans, performed at a maximum of 1 year before the reading, during two reading sessions, with an interval of 15 days, in october and november 2022
  presence of signal hyperintensity within the tendon on MRI ZTE sequence

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Norenberg D, Ebersberger HU, Walter T, Ockert B, Knobloch G, Diederichs G, Hamm B, Makowski MR. Diagnosis of Calcific Tendonitis of the Rotator Cuff by Using Susceptibility-weighted MR Imaging. Radiology. 2016 Feb;278(2):475-84. doi: 10.1148/radiol.2015150034. Epub 2015 Sep 3. PMID 26347995
- [Background] Aydingoz U, Yildiz AE, Ergen FB. Zero Echo Time Musculoskeletal MRI: Technique, Optimization, Applications, and Pitfalls. Radiographics. 2022 Sep-Oct;42(5):1398-1414. doi: 10.1148/rg.220029. Epub 2022 Jul 29. PMID 35904982